CLINICAL TRIAL: NCT01486017
Title: A Phase 1, Single-Dose, Open-Label, 3-Period, Randomized Crossover Study to Assess the Relative Bioavailability Across Three Strengths of a New ASP015K Tablet Formulation in Healthy Volunteers
Brief Title: A Single Oral Dose Study of ASP015K in Healthy Volunteers Assessing the Relative Bioavailability Across Three Tablet Strengths From a New Formulation of ASP015K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 015K-CL-PK18
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Bioavailability of ASP015K; Pharmacokinetics of ASP015K; Healthy Subjects
Keywords: ASP015K; healthy subjects; bioavailability; rheumatoid arthritis; psoriasis; transplantation
MeSH Terms: conditions — Arthritis, Rheumatoid; Psoriasis | interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): ASP015K oral dose low strength
  Interventions: Drug: ASP015K
- Treatment B (Experimental): ASP015K oral dose medium strength
  Interventions: Drug: ASP015K
- Treatment C (Experimental): ASP015K oral dose high strength
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — oral

SUMMARY:
The purpose of this study is to determine the relative bioavailability and pharmacokinetic profiles from three strengths of a new tablet formulation of ASP015K and to evaluate the safety and tolerability after a single dose of three different strengths of a new tablet formulation.

DETAILED DESCRIPTION:
Eligible subjects will be admitted on Day-1 and remain confined on the unit for 16 days. Each subject will receive a single dose of study drug per the defined treatment periods on the mornings of Day 1, Day 6 and Day11. There will be a minimum of 5 days between each consecutive dose group. Any subject discontinuing the study prior to completion should have all end of study evaluations completed.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs at least 45 kg and has a body mass index (BMI) of 18-32 kg/m2
* Male subject agrees to sexual abstinence, is surgically sterile or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method until 90 days after the last dose of study drug administration
* Male subject agrees to not donate sperm until 90 days after the dose of study drug administration
* Female subject is surgically sterile or is post-menopausal and is not pregnant and is not lactating
* Subject's 12-lead electrocardiogram (ECG) is normal
* Subject must be capable of swallowing multiple tablets

Exclusion Criteria:

* Subject has a previous history of any clinically significant gastro-intestinal, neurological, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, malignancy excluding non-melanoma skin cancer or any other medical condition
* Subject has had major GI surgery (such as colectomy, cholecystectomy, etc)
* Subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/ substance abuse within past 2 years
* Subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week
* Subject has a positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody
* Subject has a history of the human immunodeficiency virus (HIV) antibody
* Subject has a positive tuberculosis (TB) skin test, Quantiferon Gold test or T-SPOT® test
* Subject received any vaccine within 60 days
* Subject received an experimental agent within 30 days
* Subject has an absolute neutrophil count (ANC) < 2500 cells/mm3
* Subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days
* Subject has a history of smoking or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic parameters of ASP015K: Cmax, AUClast, and AUCinf | Up to Day 15

SECONDARY OUTCOMES:
Composite of pharmacokinetic parameters of ASP015K: tmax, apparent terminal elimination half-life (t1/2), apparent body clearance after oral dosing (CL/F), and apparent volume of distribution (Vz/F) | Up to Day 15
Composite of pharmacokinetic parameters of ASP015K metabolite H2: Cmax, AUClast, AUCinf, tmax and t1/2 | Up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Covance, Dallas, Texas, United States